CLINICAL TRIAL: NCT07334392
Title: Effectiveness of an Innovative Therapeutic Exercise Program on Physical and Cognitive Function in Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Impact of a Multicomponent Exercise Program on Cognitive and Functional Outcomes in Patients With Mild Cognitive Impairment
Acronym: MExeProMCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Collaborators: General University Hospital of Patras (Other); Andreas Mentzelopoulos Foundation (Unknown)
Responsible Party: Principal Investigator, Eftychia Nastou, PhD candidate, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17335/01-06-2025
Record Dates: First submitted 2025-08-21; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment; Walking; Balance; Cognition
Keywords: kinetic and kinematic; balance; global cognition; executive function; attention; mci; multicomponent program; exercise; dual tasking
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with Two Experimental Groups and one Control Group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Innovative therapeutic exercise program emphasizing in dual tasking (Experimental): Participants will perform aerobic exercises, strengthening exercises and balance exercises combined with cognitive exercises at the same time for 60- 90 minutes/ twice a week/ three months.
  Interventions: Other: Innovative therapeutic exercise program
- Therapeutic exercise program (Active Comparator): Participants will perform aerobic exercises, strengthening exercises and balance exercises for 60- 90 minutes/ twice a week/ three months.
  Interventions: Other: Therapeutic exercise program
- Control group (Active Comparator): The control group will be provided with educational material in the form of a flyer outlining the health benefits of exercise and general lifestyle recommendations.
  Interventions: Other: Flyer

INTERVENTIONS:
Other: Innovative therapeutic exercise program — Aerobic, strengthening and balance exercises combined with cognitive training -name: Experimental group 1 (EXP1)
  Arms: Innovative therapeutic exercise program emphasizing in dual tasking
Other: Therapeutic exercise program — Aerobic, strengthening and balance exercises without cognitive training- name: Experimental group 2 (EXP2)
  Arms: Therapeutic exercise program
Other: Flyer — The control group will receive only educational material in the form of a flyer, outlining the importance and potential benefits of physical activity, along with general lifestyle recommendations, without participating in the structured exercise intervention- name: Control group (CG)
  Arms: Control group

SUMMARY:
The goal of this randomised clinical trial is to investigate the effectiveness of an innovative therapeutic exercise program emphasizing in dual-task exercises in people with amnestic Mild Cognitive Impairment. The main questions it aims to answer are:

Does the innovative therapeutic exercise program improve gait and balance? Does the innovative therapeutic exercise program improve cognition?

Researchers will compare the innovative therapeutic exercise program emphasizing in dual-task exercises to a therapeutic exercise program without emphasizing in dual-task exercises and to a control group (given instruction about the benefits of exercise).

Participants will:

* Perform the exercise program twice a week for three months.
* Will be assessed before and after the intervention.
* Will record The Borg Scale of Perceived Exertion every second week to monitor and assess the progression of exercise intensity.

ELIGIBILITY:
Inclusion Criteria:

* individuals > 50 years old
* people with confirmed cognitive impairment, as evidenced by values within normal limits on the Montreal Cognitive Assessment test (MOCA ) >20
* stable medication in the last month
* independent walking

Exclusion Criteria:

* people with dementia
* people suffering from chronic mental illness (e.g. schizophrenia, bipolar disorder)
* people suffering from a neurological disorder or injuries (e.g. multiple sclerosis, Parkinson's, traumatic brain injury)
* people with clinical depression (as determined by the Neuropsychiatric Inventory (NPI) assessment and medical diagnosis)
* people who have had recent surgery
* people with insufficient knowledge of the Greek language

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Kinematic and kinetic gait assessment | baseline, post- intervention (12 weeks)
  Participants will be instructed to walk at their self-selected, comfortable walking pace. Gait performance will be assessed under four task conditions: single-task walking, dual-task walking, single-task obstacle crossing, and dual-task obstacle crossing. These conditions are designed to evaluate participants' walking ability and adaptability under both simple and cognitively demanding circumstances.
  Duration: ≈ 40 minutes
Functional Gait Assessment (FGA) | baseline, post- intervention (12 weeks)
  The Functional Gait Assessment is a clinical tool used to evaluate postural stability during various walking tasks. The assessment includes 10 standardized walking tasks, each addressing a distinct aspect of gait and balance. Performance on each task is rated on a 4-point ordinal scale (0-3), where higher scores indicate better functional performance. The total score ranges from 0 to 30, with a higher total score representing normal gait and balance, and a lower score indicating gait instability or impaired functional mobility.
  Test duration: ≈ 10-15 minutes
mini Balance Evaluation Systems Test (mini-BESTest) | baseline, post- intervention (12 weeks)
  The Mini-BESTest is a clinical balance assessment tool designed to evaluate dynamic balance control and identify the specific balance systems affected in individuals with balance disorders. It is a shortened version of the original Balance Evaluation Systems Test (BESTest).
  It comprises 14 items, each scored on a 3-point ordinal scale (0-2), with a maximum total score of 28 points.
  The assessment includes four subscales, each representing a specific component of balance control:
  Anticipatory Postural Adjustments - maximum score: 6 points Reactive Postural Control - maximum score: 6 points Sensory Orientation - maximum score: 6 points Dynamic Gait - maximum score: 10 points Higher scores indicate better balance performance, while lower scores reflect greater balance impairment.
  Test duration: ≈ 15minutes
Montreal Cognitive Assessment (MoCA) | baseline, post- intervention (12 weeks)
  The MoCA assesses global cognitive function across multiple domains. It includes 12 brief tasks, grouped into 7 cognitive domains:
  Total possible score: 30 points. Each task contributes a set number of points according to its complexity. If the individual has ≤ 12 years of education, 1 additional point is added to the total score to account for educational effects.
  Higher score indicates better global cognition while lower scores indicate impairment Administration time: ≈ 10-15 minutes
Cognitive Telephone Screening Instrument (COGTEL) | baseline, post- intervention (12 weeks)
  The test consists of six subtests, each targeting a specific cognitive domain:
  1. Prospective Memory:(Score range: 0-2 points)
  2. Verbal Short-Term Memory: (Score range: 0-8 points)
  3. Verbal Long-Term Memory : (Score range: 0-8 points)
  4. Working Memory (Backward Digit Span): (Score range: 0-12 points)
  5. Verbal Fluency: (Score = number of correct words produced)
  6. Inductive Reasoning: (Score range: 0-8 points)
  Each subtest yields an individual score, which are combined into a total composite score using a weighted formula reflecting the relative contribution of each domain to overall cognition:
  Total COGTEL score =(7.2 × Prospective Memory) + (1.0 × Verbal Short-Term Memory) + (0.9 × Verbal Long-Term Memory) + (0.8 × Working Memory) + (0.2 × Verbal Fluency) + (1.7 × Inductive Reasoning) Higher score indicates better cognitive performance while lower scores indicate impairment Administration time: ≈ 10-15 minutes
Stroop Test | baseline, post- intervention (12 weeks)
  The Stroop test is a sensitive index of executive function and attention. During the task, the participant is required to name the color of the ink in which a word is printed rather than read the word itself.
  Total number of correct responses within a set time limit (60 seconds), and number of errors (including self-corrections and uncorrected errors) are calculated.
  Higher scores indicate better executive control, while lower or negative scores suggest difficulty inhibiting automatic responses.
  Administration time: ≈5-10 minutes

SECONDARY OUTCOMES:
Lipid profile | baseline, post- intervention (12 weeks)
  Plasma samples will be collected from the participants and will be analyzed using standardized biochemical and immunoassay techniques. The samples will be analyzed to assess changes associated with the intervention.
  Parameters Measured: total cholesterol Blood sample collection: ≈ 5 minutes
Hand grip strength test | baseline, post- intervention (12 weeks)
  The Hand Grip Strength Test is a widely used assessment of upper limb muscle strength, particularly of the forearm and hand flexor muscles. The test measures maximum isometric grip force, which reflects not only upper limb strength but also overall muscle function.The participant holds the dynamometer and squeezes as hard as possible for 3-5 seconds. Three trials are performed per hand, with 30-60 seconds of rest between trials. The mean score of the three trials (kg) are reported for each hand. Results are compared to age- and sex-specific normative data.
  Administration time: ≈ 3- 5 minutes
30 Second Sit to Stand Test | baseline, post- intervention (12 weeks)
  The 30-Second Sit-to-Stand Test (also known as the 30-Second Chair Stand Test) is a simple, reliable measure of lower limb strength, endurance, and functional mobility. Participant sits in the middle of the chair, back straight, feet flat on the floor, shoulder-width apart, and arms crossed over the chest. On the command "Go," the participant stands up fully and sits down as many times as possible within 30 seconds. The participant must fully extend the knees and hips when standing and sit back fully each time. Partial stands do not count. The assessor counts the number of completed stands within 30 seconds. More repetitions indicate better lower-body strength and endurance. Scores below age- and sex-specific norms indicate reduced lower-body strength and increased fall risk.
  Administration time: ≈2-3 minutes
Falls Efficacy Scale - International (FES-I) | baseline, post- intervention (12 weeks)
  The Falls Efficacy Scale - International (FES-I) is a standardized self-report questionnaire designed to assess an individual's concern or fear of falling during various everyday activities. The original FES-I includes 16 items, each describing a common daily activity. Participants rate their concern about falling while performing each activity, regardless of whether they actually do it. Each item is rated on a 4-point Likert scale: 1 (Not at all concerned)-4 (Very concerned). Total Score: 16-64 points. Higher scores indicate greater concern about falling and lower confidence in performing activities safely.
  Administration time: ≈10 minutes
6 Minute Walk Test (6MWT) | baseline, post- intervention (12 weeks)
  The 6-Minute Walk Test is a widely used test to assess functional exercise capacity. It measures the distance an individual can walk on a flat, hard surface in six minutes. The participant is instructed to walk as far as possible for 6 minutes, at their own pace, without running. They may slow down, stop, and rest if necessary, but should resume walking as soon as they are able. Standardized encouragements are given at each minute (e.g., "You are doing well. Keep up the good work"). The total distance walked in meters is recorded at the end of 6 minutes.
  Total administration time: ≈ 10-15 minutes (including preparation and recovery)
Timed Up and Go test (TUG) | baseline, post- intervention (12 weeks)
  The TUG test measures functional mobility, specifically the time it takes for a person to rise from a chair, walk a short distance, turn, return, and sit down again. The participant begins seated in a standard armchair (seat height ≈ 45 cm).
  On the command "Go," the participant must: Stand up from the chair,Walk 3 meters (10 feet) at a comfortable and safe pace,Turn around,Walk back to the chair, and sit down again.The timer starts when the participant's back leaves the chair and stops when they sit down again. Lower times indicate better functional mobility. Higher times suggest mobility impairment and increased fall risk.
  Test duration: ≈ 3-5 minutes
Short Physical Performance Battery- (SPPB) | baseline, post- intervention (12 weeks)
  The Short Physical Performance Battery (SPPB) is a standardized test used to assess lower extremity function, mobility, and physical performance in older adults. The SPPB consists of three main components, each assessing a different aspect of lower-body performance: Standing Balance Test, Gait Speed Test, Chair Stand Test. Each of the three components is scored on a 0-4 scale, based on performance time or ability. Component scores (0-4) are summed to give a total score (0-12). Higher scores indicate better functional performance, while lower scores reflect greater functional limitation.
  Test duration: ≈ 10minutes
Exercise Adherence Rating Scale (EARS) | end of 4 weeks of intervention, end of 8 weeks of intervention, end of intervention (12 weeks)
  The EARS is a self-report questionnaire designed to measure how well individuals adhere to prescribed exercise programs. The EARS comprises three sections (A, B, and C) though the primary adherence measurement is in Section B.
  Section A: Captures qualitative information about the prescribed exercise (type, frequency) as given by the healthcare provider.
  Section B: Contains 6 items that assess exercise adherence behavior. Section C: Contains 10 items related to reasons for non-adherence (barriers and facilitators).
  The 6 adherence items of Section B are each scored on a 5-point Likert scale: 0 = "strongly agree" to 4 = "strongly disagree".
  The sum of the 6 items yields a raw adherence score ranging from 0 to 24. A higher score indicates better adherence to the prescribed exercise protocol. Total administration time (including instructions): ≈5 minutes
Word Finding Questionnaire - Brief Version (WoFi-Brief) | baseline, post- intervention (12 weeks)
  The WoFi-Brief is a shortened version of the WoFi (Word Finding) questionnaire, which is used to assess difficulties in word retrieval. The WoFi-Brief consists of 16 items and is designed to efficiently evaluate an individual's word-finding ability. Each item is rated on a Likert-type scale that reflects the frequency or severity of word-finding problems. Scores are summed to yield a total score, with higher scores indicating greater perceived word-finding difficulty.
  Administration time: ≈5 minutes
Consortium to Establish a Registry for Alzheimer's Disease-CERAD constructional praxis (CP) and constructional praxis recall | baseline, post- intervention (12 weeks)
  Consortium to Establish a Registry for Alzheimer's Disease- CERAD constructional praxis (CP) and constructional praxis recall are subtests of the CERAD neuropsychological battery designed to assess visuospatial abilities and memory. The CP copying task involves the patient copying 4 geometric figures, while the CP recall task assesses the patient's ability to remember and reproduce these same figures after a delay. Performance is scored on an 11-point scale based on standardized criteria evaluating the accuracy, proportionality, spatial organization, and completeness of each drawing. Higher scores indicate better visuospatial performance.
  Administration time: ≈5-10 minutes
Geriatric Depression Scale - 15 Item Version | baseline, post- intervention (12 weeks)
  The Geriatric Depression Scale, 15-item version (GDS-15), is a widely used self-report screening instrument designed to assess depressive symptoms in older adults. It consists of 15 yes/no items that evaluate mood, motivation, energy, and cognitive-emotional symptoms associated with depression. Scoring is conducted by assigning 1 point to each response indicative of depressive symptomatology, resulting in a total score that ranges from 0 to 15.Higher scores indicate greater severity of depressive symptomatology.
  Administration time: ≈5 minutes
The Neuropsychiatric Inventory-12 Item Version | baseline, post- intervention (12 weeks)
  The Neuropsychiatric Inventory-12 (NPI-12) is a structured, informant-based assessment designed to measure the presence and severity of behavioral and psychological symptoms in individuals with neurocognitive disorders. The instrument evaluates 12 neuropsychiatric domains: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep disturbances, and appetite/eating changes. For each domain endorsed, the informant rates frequency (1-4) and severity (1-3). The domain score is calculated by multiplying frequency and severity, yielding values from 1 to 12 per domain. A separate caregiver distress rating (0-5) is also obtained for each domain to quantify the emotional impact on the caregiver. Total NPI-12 scores are derived by summing all domain scores, with higher scores reflecting greater neuropsychiatric symptom burden.
  Administration time: ≈10 to 20 minutes

OTHER OUTCOMES:
Weekly diaries | throughout the intervention (12 weeks)
  Exercise providers will complete a weekly attendance and performance log for each participant enrolled in the exercise program. The log will document participant attendance, exercise compliance, and qualitative feedback on performance. This information will be used to progressively adjust the difficulty level of the exercises Duration: ≈ 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, University of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Yes
happy to share the results after after processing all the data